CLINICAL TRIAL: NCT01349959
Title: Phase II Study of Azacitidine and Entinostat (SNDX-275) in Patients With Advanced Breast Cancer
Brief Title: Azacitidine and Entinostat in Treating Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02585; NCI-2011-02585 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000698726; SKCCC J1107 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 8822 (Other: CTEP); N01CM00099 (NIH); N01CM00038 (NIH); N01CM62205 (NIH); P30CA006973 (NIH); U01CA099168 (NIH); U01CA070095 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Male Breast Carcinoma; Recurrent Breast Carcinoma; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Azacitidine; entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (entinostat and azacitidine) (Experimental): Patients receive azacitidine SC on days 1-5 and 8-10, and entinostat PO on days 3 and 10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may continue azacitidine and entinostat in combination with hormonal therapy, at treating physician discretion, or undergo event monitoring.
  Interventions: Drug: Azacitidine; Drug: Entinostat; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS 275; MS-275; MS275; SNDX 275; SNDX-275; SNDX275
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well giving azacitidine and entinostat work in treating patients with advanced breast cancer. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Entinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving azacitidine together with entinostat may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate objective response rate by Response Evaluation Criteria In Solid Tumors (RECIST) criteria of the combination of azacitidine (5-AZA) and entinostat in women with advanced breast cancer; triple-negative and hormone-refractory.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of the combination of 5-AZA and entinostat in women with advanced breast cancer.

II. To determine progression-free survival, overall survival, and clinical benefit rate of the combination of 5-AZA and entinostat.

TERTIARY OBJECTIVES:

I. To collect safety and toxicity data as well as the feasibility and response rate where hormonal therapy is added to the combination under investigation at the time of progressive disease. (Exploratory) II. To determine the pharmacokinetic profile of 5-AZA (full profile) and entinostat (trough concentrations) in patients with advanced breast cancer. (Exploratory) III. To assess serum cytidine deaminase pharmacogenetics and phenotypic activity as a potential biomarker of response to 5-AZA. (Exploratory) IV. To evaluate baseline and change in candidate gene re-expression (e.g., estrogen receptor [ER] alpha, retinoic acid receptor [RAR] beta) in malignant tissue obtained from selected patients through fine-needle aspiration (FNA) and core biopsy, prior to and following combination therapy. (Exploratory) V. To evaluate baseline and change in gene methylation silencing in circulating deoxyribonucleic acid (DNA) obtained prior to and following combination therapy. (Exploratory) VI. To evaluate baseline and change in gene methylation in malignant tissue obtained through FNA and core biopsy. (Exploratory)

OUTLINE: This is a multicenter study.

Patients receive azacitidine subcutaneously (SC) on days 1-5 and 8-10, and entinostat orally (PO) on days 3 and 10. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may continue azacitidine and entinostat in combination with hormonal therapy, at treating physician discretion, or undergo event monitoring.

After completion of study therapy, patients are followed up every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed adenocarcinoma of the breast triple-negative (ER-, progesterone receptor [PR]-, human epidermal growth factor receptor 2 [HER2]-) or hormone positive/ HER2-, with evidence of locally advanced and inoperable or metastatic disease (American Joint Committee on Cancer [AJCC] Stage IV)

  * NOTE: Triple-negative patients will be defined per American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) Guidelines; these guidelines state that ER and PR assays be considered positive if there are at least 1% positive tumor nuclei in the sample on testing in the presence of expected reactivity of internal (normal epithelial elements) and external controls
  * A patient who has a change in receptor status (e.g., PR negative to positive) may be stratified as triple negative or hormone positive, contrary to the most recent receptor testing, for the purposes of the study based upon the clinical course at the discretion of the Study Chair; for HER2 assessment, a negative result is an immuno-histochemistry staining of 0 or 1+, a fluorescence in situ hybridization (FISH) result of less than 4.0 HER2 gene copies per nucleus, or a FISH ratio of less than 1.8
* Patients with triple negative disease must have progressed through at least 1 prior chemotherapy regimen (administered in the adjuvant or metastatic setting); hormone receptor-positive patients must have progressed through two lines of hormonal therapy (administered in the adjuvant or metastatic setting), unless otherwise eligible as per below, and at least 1 prior chemotherapy regimen (administered in the adjuvant or metastatic setting) with no known curative options available

  * NOTE: Patients with hormone receptor-positive disease may be considered eligible if deemed clinically hormone-resistant taking into consideration the rate of progression of disease or a short interval of time on first line hormonal therapy before progression, or if intolerant of hormonal therapy such that further hormonal therapy will not be considered as part of the treatment strategy
* In patients with metastatic disease in the liver, liver disease burden is limited to no more than 30% of total liver volume as assessed by local review
* Patients must have measurable disease
* Life expectancy of >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Hemoglobin (HgB) >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN); an exception to this may be allowed for participants with Gilbert's syndrome with documented approval by the Protocol Chair
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x ULN
* Creatinine =< institutional ULN or creatinine clearance >= 60 mL/min using the Modified Cockcroft-Gault formula
* Negative (serum or urine) pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Patient must have an accessible tumor lesion from which a biopsy specimen can be obtained; NOTE: if baseline biopsy is attempted and is unsuccessful (eg, patient intolerance, inadequate tissue), the patient will still be considered eligible for the study
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to provide tissue and blood samples for mandatory translational research
* Willingness to return to the enrolling institution for follow-up

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
  * NOTE: should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Any of the following:

  * Chemotherapy < 3 weeks prior to registration
  * Hormone therapy < 3 weeks prior to registration
  * Radiotherapy < 3 weeks prior to registration
  * Surgery < 3 weeks prior to registration
  * Nitrosoureas/mitomycin C < 6 weeks prior to registration
  * Trastuzumab < 6 weeks prior to registration
  * Bevacizumab < 6 weeks prior to registration
  * Those who have not recovered from acute adverse events to grade < 2 or baseline due to agents administered, with exception of alopecia, unless approved by the Protocol Chair
  * NOTE: concurrent bisphosphonate therapy is allowed; concurrent ovarian suppression therapy (i.e., Lupron or Zoladex) is also allowed at the discretion of the Protocol Chair/designee
* Any other ongoing investigational agents
* Known sensitivity to 5-AZA, entinostat or mannitol
* Uncontrolled intercurrent illness that in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure (New York Heart Association [NYHA] class II or above)
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Other co-morbid systemic illness or other severe concurrent disease
* Active malignancy other than breast cancer =< 3 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Received prior treatment with HDAC (histone deacetylase) inhibitors or demethylating agents =< 2 weeks prior to registration
* Unstable brain metastases; NOTE: patients with brain metastases must have stable neurologic status and magnetic resonance imaging (MRI) imaging following local therapy (surgery or radiation) for at least 4 weeks, with no dexamethasone requirement (stable low dose dexamethasone allowed at discretion of Study Chair); patients with leptomeningeal disease are not eligible
* Patient taking valproic acid
* Patient who cannot swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2014-03-27 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Unity Hospital, Fridley, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Li H, Chiappinelli KB, Guzzetta AA, Easwaran H, Yen RW, Vatapalli R, Topper MJ, Luo J, Connolly RM, Azad NS, Stearns V, Pardoll DM, Davidson N, Jones PA, Slamon DJ, Baylin SB, Zahnow CA, Ahuja N. Immune regulation by low doses of the DNA methyltransferase inhibitor 5-azacitidine in common human epithelial cancers. Oncotarget. 2014 Feb 15;5(3):587-98. doi: 10.18632/oncotarget.1782. PMID 24583822

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 58 consented, 18 screen failed and did not receive study treatment
Period: Overall Study
Arm/Group | Treatment (Entinostat and Azacitidine)
Started | 40
Completed | 33
Not Completed | 7
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 31
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (Percentage of Participants With Complete or Partial Response Noted as the Objective Status on Two Consecutive Evaluations at Least 4 Weeks Apart) Assessed by RECIST
Description: Percentage of participants with complete or partial response will be estimated independently for each cohort by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: Up to 3 years
Population: There were 13/40 participants with triple-negative breast cancer (TNBC) and 27/40 participants with hormone-resistant breast cancer (HRBC).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 40
percentage of participants
  Triple-negative Breast Cancer (TNBC): number analyzed (Participants) | 13
  Triple-negative Breast Cancer (TNBC) | 0 [NA to NA] — No clinical response was observed in participants with TNBC.
  Hormone-resistant Breast Cancer (HRBC): number analyzed (Participants) | 27
  Hormone-resistant Breast Cancer (HRBC) | 4 [0 to 19]

2. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate estimated by the number of patients who achieve a confirmed response plus the number of patients who have stable disease for a duration of at least 6 months divided by the total number of evaluable patients. All evaluable patients will be used for this analysis.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 40
Participants
  TNBC: number analyzed (Participants) | 13
  TNBC | 0
  HRBC: number analyzed (Participants) | 27
  HRBC | 1

3. Secondary Outcome: Overall Survival
Description: Median number of months alive, estimated by Kaplan-Meier method.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 40
months
  TNBC: number analyzed (Participants) | 13
  TNBC | 6.6 [2.0 to 10.3]
  HRBC: number analyzed (Participants) | 27
  HRBC | 12.6 [6.3 to 16.3]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Median number of months without progression. Estimated using the method of Kaplan-Meier.
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 40
months
  TNBC: number analyzed (Participants) | 13
  TNBC | 1.4 [0.9 to 1.8]
  HRBC: number analyzed (Participants) | 27
  HRBC | 1.8 [1.7 to 1.9]

5. Other Pre Specified Outcome: Number of Participants With Change in Expression of Relevant Genes (e.g., ER Alpha and RAR Beta) Evaluated by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)
Description: Number of participants with a change in candidate gene re-expression of ER-alpha and RAR beta evaluated by reverse transcriptase polymerase chain reaction (RT-PCR).
Time Frame: Baseline to up to 8 weeks
Population: There were 13/40 participants with triple-negative breast cancer (TNBC) and 27/40 participants with hormone-resistant breast cancer (HRBC). However, data was only evaluable in 19/40 participants (5/13 TNBC, and 14/40 HRBC).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 19
Participants
  TNBC: number analyzed (Participants) | 5
  TNBC | 0
  HRBC: number analyzed (Participants) | 14
  HRBC | 14

6. Other Pre Specified Outcome: Circulating DNA Evaluated Using QM-MSP
Description: Data will also be graphically displayed showing trend in median values across time. Nonparametric Wilcoxon signed rank tests will be used to determine whether or not the data shows evidence of changes from baseline.
Time Frame: Up to 8 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Confirmed Response Rate to Azacitidine and Entinostat Plus the Addition of Hormone Therapy
Description: Will be estimated in each cohort. All evaluable patients who receive hormonal therapy will be used for this analysis.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 40
Participants
  TNBC: number analyzed (Participants) | 13
  TNBC | 0
  HRBC: number analyzed (Participants) | 27
  HRBC | 1

8. Other Pre Specified Outcome: Feasibility of the Addition of Hormone Therapy, Evaluated by Calculating the Number of Patients With Disease Progression That go on to Receive Hormonal Therapy
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 40
Participants
  TNBC: number analyzed (Participants) | 13
  TNBC | 4
  HRBC: number analyzed (Participants) | 27
  HRBC | 12

9. Other Pre Specified Outcome: Number of Participants With Change in Gene Methylation Evaluated Using Quantitative Multiple Methylation-specific Polymerase Chain Reaction (QM-MSP)
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Entinostat and Azacitidine)
Number analyzed (Participants) | 40
Participants
  TNBC: number analyzed (Participants) | 13
  TNBC | 0
  HRBC: number analyzed (Participants) | 27
  HRBC | 14

ADVERSE EVENTS:
Time Frame: 1 year
Description: CTCAE criteria
Arm/Group | Treatment (Entinostat and Azacitidine)
All-Cause Mortality (participants affected / at risk) | 33/40
Serious Adverse Events (participants affected / at risk) | 2/40
Other Adverse Events (participants affected / at risk) | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Entinostat and Azacitidine) (N=40)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Death (General disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Entinostat and Azacitidine) (N=40)
Neutropenia (Blood and lymphatic system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less